CLINICAL TRIAL: NCT05067166
Title: Open-Label, Expanded Access Protocol of a Human Monoclonal Antibody, Ansuvimab (mAb114), Administered As a Therapeutic to Ebola-Infected Patients or As a High-Risk Ebola Post-Exposure Prophylaxis
Brief Title: Open-Label Expanded Access for Ebola-Infected Patients to Receive Human MAb Ansuvimab As Therapeutic or for HR PEP
Status: Available | Type: Expanded Access
Sponsor: Ridgeback Biotherapeutics, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: Ansuvimab EAP
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Ebola Virus Disease
Keywords: EBANGA; orthoebolavirus zairense, EBOV; ansuvimab; Zaire ebolavirus, EVD; Compassionate Use; Ebola
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — ansuvimab

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: Ansuvimab — single infusion 50 mg/kg IV
  Other Names: mAb114, Ebanga

SUMMARY:
The human monoclonal antibody (mAb), ansuvimab (mAb114), will be provided to Ebola-infected patients as either a treatment or as PEP under an expanded access protocol. Ansuvimab is administered at 50 mg/kg as a single intravenous (IV) infusion

DETAILED DESCRIPTION:
This is an open-label, intermediate-size patient population, expanded access protocol (EAP) of ansuvimab administered once by IV infusion at a dose of about 50 mg/kg (weight-based dosing). Participants will be monitored and assessed daily for safety, including clinical observation, laboratory monitoring, the incidence of adverse events (AEs) and serious adverse events (SAEs) as defined by protocol, including AEs that by clinical judgement are atypical for orthoebolavirus zairense (EBOV) in infected patients, and any AEs that occur during product infusions. PEP participants will be followed to determine outcome following ansuvimab administrations through the study period for EBOV status (positive/negative). Blood will be collected for protocol-specific assessments and RT-PCR evaluation of viral load by available assay. A blood sample for Ebolavirus viral load measurement will be collected before mAb114 administration and at subsequent study time points per the Schedule of Evaluations. Participants will be followed for a period as defined by protocol after the product administration. Survival status for infected patients and follow up for PEP participants for signs/symptoms of EBOV will be recorded as applicable.

Ansuvimab will be provided for expanded access in any EBOV outbreak location as authorized by the applicable Regulatory Authorities and/or Ethics Committee(s).

ELIGIBILITY:
Inclusion Criteria:

* Male or female with laboratory confirmed (based on local standard of care) EBOV infection or with recent high-risk EBOV exposure as determined by a treating Physician or designee.
* Able to provide proof of identity to the satisfaction of the clinical team
* Able and willing to complete the informed consent process personally, or if the patient is unable to do so, then informed consent completed by a legally-authorized representative according to local laws and regulations.

Exclusion Criteria:

- Any medical condition that, in the opinion of the Treating Physician, would place the patient at an unreasonably increased risk through participation in this treatment protocol.

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Background] Bebell LM, Riley LE. Ebola virus disease and Marburg disease in pregnancy: a review and management considerations for filovirus infection. Obstet Gynecol. 2015 Jun;125(6):1293-1298. doi: 10.1097/AOG.0000000000000853. PMID 26000499
- [Background] Broadhurst MJ, Brooks TJ, Pollock NR. Diagnosis of Ebola Virus Disease: Past, Present, and Future. Clin Microbiol Rev. 2016 Oct;29(4):773-93. doi: 10.1128/CMR.00003-16. PMID 27413095
- [Background] Cherif MS, Koonrungsesomboon N, Kasse D, Cisse SD, Diallo SB, Cherif F, Camara F, Kone A, Avenido EF, Diakite M, Diallo MP, Le Gall E, Cisse M, Karbwang J, Hirayama K. Ebola virus disease in children during the 2014-2015 epidemic in Guinea: a nationwide cohort study. Eur J Pediatr. 2017 Jun;176(6):791-796. doi: 10.1007/s00431-017-2914-z. Epub 2017 Apr 25. PMID 28444452
- [Background] Corti D, Misasi J, Mulangu S, Stanley DA, Kanekiyo M, Wollen S, Ploquin A, Doria-Rose NA, Staupe RP, Bailey M, Shi W, Choe M, Marcus H, Thompson EA, Cagigi A, Silacci C, Fernandez-Rodriguez B, Perez L, Sallusto F, Vanzetta F, Agatic G, Cameroni E, Kisalu N, Gordon I, Ledgerwood JE, Mascola JR, Graham BS, Muyembe-Tamfun JJ, Trefry JC, Lanzavecchia A, Sullivan NJ. Protective monotherapy against lethal Ebola virus infection by a potently neutralizing antibody. Science. 2016 Mar 18;351(6279):1339-42. doi: 10.1126/science.aad5224. Epub 2016 Feb 25. PMID 26917593
- [Background] Fischer WA 2nd, Vetter P, Bausch DG, Burgess T, Davey RT Jr, Fowler R, Hayden FG, Jahrling PB, Kalil AC, Mayers DL, Mehta AK, Uyeki TM, Jacobs M. Ebola virus disease: an update on post-exposure prophylaxis. Lancet Infect Dis. 2018 Jun;18(6):e183-e192. doi: 10.1016/S1473-3099(17)30677-1. Epub 2017 Nov 15. PMID 29153266
- [Background] Gaudinski MR, Coates EE, Novik L, Widge A, Houser KV, Burch E, Holman LA, Gordon IJ, Chen GL, Carter C, Nason M, Sitar S, Yamshchikov G, Berkowitz N, Andrews C, Vazquez S, Laurencot C, Misasi J, Arnold F, Carlton K, Lawlor H, Gall J, Bailer RT, McDermott A, Capparelli E, Koup RA, Mascola JR, Graham BS, Sullivan NJ, Ledgerwood JE; VRC 608 Study team. Safety, tolerability, pharmacokinetics, and immunogenicity of the therapeutic monoclonal antibody mAb114 targeting Ebola virus glycoprotein (VRC 608): an open-label phase 1 study. Lancet. 2019 Mar 2;393(10174):889-898. doi: 10.1016/S0140-6736(19)30036-4. Epub 2019 Jan 24. PMID 30686586
- [Background] Jacobs M, Aarons E, Bhagani S, Buchanan R, Cropley I, Hopkins S, Lester R, Martin D, Marshall N, Mepham S, Warren S, Rodger A. Post-exposure prophylaxis against Ebola virus disease with experimental antiviral agents: a case-series of health-care workers. Lancet Infect Dis. 2015 Nov;15(11):1300-4. doi: 10.1016/S1473-3099(15)00228-5. Epub 2015 Aug 25. PMID 26321189
- [Background] Mbala-Kingebeni P, Aziza A, Di Paola N, Wiley MR, Makiala-Mandanda S, Caviness K, Pratt CB, Ladner JT, Kugelman JR, Prieto K, Chitty JA, Larson PA, Beitzel B, Ayouba A, Vidal N, Karhemere S, Diop M, Diagne MM, Faye M, Faye O, Aruna A, Nsio J, Mulangu F, Mukadi D, Mukadi P, Kombe J, Mulumba A, Villabona-Arenas CJ, Pukuta E, Gonzalez J, Bartlett ML, Sozhamannan S, Gross SM, Schroth GP, Tim R, Zhao JJ, Kuhn JH, Diallo B, Yao M, Fall IS, Ndjoloko B, Mossoko M, Lacroix A, Delaporte E, Sanchez-Lockhart M, Sall AA, Muyembe-Tamfum JJ, Peeters M, Palacios G, Ahuka-Mundeke S. Medical countermeasures during the 2018 Ebola virus disease outbreak in the North Kivu and Ituri Provinces of the Democratic Republic of the Congo: a rapid genomic assessment. Lancet Infect Dis. 2019 Jun;19(6):648-657. doi: 10.1016/S1473-3099(19)30118-5. Epub 2019 Apr 15. PMID 31000464
- [Background] Misasi J, Gilman MS, Kanekiyo M, Gui M, Cagigi A, Mulangu S, Corti D, Ledgerwood JE, Lanzavecchia A, Cunningham J, Muyembe-Tamfun JJ, Baxa U, Graham BS, Xiang Y, Sullivan NJ, McLellan JS. Structural and molecular basis for Ebola virus neutralization by protective human antibodies. Science. 2016 Mar 18;351(6279):1343-6. doi: 10.1126/science.aad6117. Epub 2016 Feb 25. PMID 26917592
- [Background] Moekotte AL, Huson MA, van der Ende AJ, Agnandji ST, Huizenga E, Goorhuis A, Grobusch MP. Monoclonal antibodies for the treatment of Ebola virus disease. Expert Opin Investig Drugs. 2016 Nov;25(11):1325-1335. doi: 10.1080/13543784.2016.1240785. Epub 2016 Oct 8. PMID 27676206
- [Background] Sullivan N, Yang ZY, Nabel GJ. Ebola virus pathogenesis: implications for vaccines and therapies. J Virol. 2003 Sep;77(18):9733-7. doi: 10.1128/jvi.77.18.9733-9737.2003. No abstract available. PMID 12941881
- See also: Ridgeback Biotherapeutics (corporate website) — http://www.ridgebackbio.com
- See also: WHO: Guidance for managing ethical issues in infectious disease outbreaks — https://apps.who.int/iris/handle/10665/250580
- See also: WHO: Notes for the record: Consultation on Monitored Emergency Use of Unregistered and Investigational Interventions for Ebola Virus Disease (EVD) — https://www.who.int/publications/m/item/consultation-on-monitored-emergency-use-of-unregistered-and-investigational-interventions-for-ebola-virus-disease